CLINICAL TRIAL: NCT04800042
Title: Study of the Prevalence of Iron Deficiency in Patients With Scheduled Major Surgery (CARENFER PBM)
Acronym: CARENFER-PBM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VIFORFRANCE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARENFER-PBM
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Diagnostic
MeSH Terms: conditions — Disease | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with scheduled major surgery (Other): Patients with scheduled major surgery
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — Blood iron status : ferritin and transferrin saturation factor

SUMMARY:
Many patients who are candidates for scheduled major surgery have a pre-operative iron deficiency which is poorly diagnosed. The management of per-operative iron deficiency is a part of the concept of the "Patient Blood Management", which is a concept recommended by health regulatory agencies in many countries. The objective of this study is to obtain updated data on the prevalence of iron deficiency in France in patients undergoing a scheduled major surgery, applying the French recommendations (determination of ferritinemia and Transferrin Saturation Factor).

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age
* Patient with scheduled major surgery
* Patient with signed consent

Exclusion Criteria:

* Protected patient : major under guardianship, tutorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood iron status | Preoperative
  Ferritin
Complete blood iron status | Preoperative
  Transferrin Saturation Factor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capdevila X, Lasocki S, Duchalais A, Rigal JC, Mertl P, Ghewy P, Farizon F, Lanz T, Buckert A, Belarbia S, Trochu JN, Cacoub P. Perioperative Iron Deficiency in Patients Scheduled for Major Elective Surgeries: A French Prospective Multicenter Cross-Sectional Study. Anesth Analg. 2023 Aug 1;137(2):322-331. doi: 10.1213/ANE.0000000000006445. Epub 2023 Mar 7. PMID 36881542